CLINICAL TRIAL: NCT00000258
Title: Role of Instructions in Nitrous Oxide Effects and Choice
Brief Title: Role of Instructions in Nitrous Oxide Effects and Choice - 10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: NIDA-08391-10; R01DA008391 (NIH); R01-08391-10
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; instruction; subjective effects; reinforcer; healthy volunteer
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Informed group (Active Comparator): Group inhaled placebo and varying doses of nitrous oxide in pairs then chose which they wanted for a third inhalation.
  Interventions: Drug: Nitrous oxide 10% & placebo; Drug: Nitrous oxide 20% & placebo; Drug: Nitrous oxide 30% & placebo; Drug: Nitrous oxide 40% and placebo
- Non-informed Group (Active Comparator): Group and technician were blinded as to which gas they were inhaling in pairs with third inhalation subject's choice.
  Interventions: Drug: Nitrous oxide 10% & placebo; Drug: Nitrous oxide 20% & placebo; Drug: Nitrous oxide 30% & placebo; Drug: Nitrous oxide 40% and placebo

INTERVENTIONS:
Drug: Nitrous oxide 10% & placebo
Drug: Nitrous oxide 20% & placebo
Drug: Nitrous oxide 30% & placebo
Drug: Nitrous oxide 40% and placebo

SUMMARY:
The purpose of this study is to conduct experiments to examine subjective and reinforcing effects of nitrous oxide. Mood altering and psychomotor effects will be tested on non-drug abusers and preference procedures will be used to assess reinforcing effects. Comparisons between nitrous oxide, opiates, and benzodiazepine antagonists will be made. To evaluate the role of instructions in nitrous oxide subjective effects and choice.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 1996-04; Primary Completion 1997-11 (Actual); Study Completion 1997-11 (Actual)

PRIMARY OUTCOMES:
Choice of nitrous oxide vs placebo | After 30 min inhalation of each
  Subjects inhaled placebo and varying per centages of nitrous oxide in sampling pair, then chose for third inhalation. One group was told which of the gases they were inhaling during sampling and one group as well as the technician administering the inhalant was blinded. Psychomotor tests were done at each dose.

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States

REFERENCES:
- [Background] Zacny JP, Cho AM, Toledano AY, Galinkin J, Coalson DW, Klock PA, Klafta JM, Young CJ. Effects of information on the reinforcing, subjective, and psychomotor effects of nitrous oxide in healthy volunteers. Drug Alcohol Depend. 1997 Nov 25;48(2):85-95. doi: 10.1016/s0376-8716(97)00114-2. PMID 9363407